CLINICAL TRIAL: NCT05231915
Title: Prevalence of the c.853delT Mutation of the HOXB13 Gene in Prostate Cancer in Martinique
Acronym: HOXB13_Mart
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 19_RIPH2_14
Record Dates: First submitted 2022-02-01; First posted 2022-02-09 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Martinique; HOXB13 c.853delT prevalence
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HOXB13 c.853delT mutation (Other): Mutation is detected using Next Generation Sequencing (NGS) technique
  Interventions: Genetic: HOXB13 c.853delT mutation

INTERVENTIONS:
Genetic: HOXB13 c.853delT mutation — Identify the Allelic frequency of the HOXB13 c.853delT mutation in patients with a cancer prostate in Martinique

SUMMARY:
In Martinique, prostate cancer incidence rates are nowadays among the highest worldwide with a high incidence of early-onset and familial forms. We identified a rare heterozygous germline variant c.853delT (p.Ter285Lysfs) rs77179853, reported only among patients of African ancestry with a minor allele frequency of 3.2%. We search to estimate the prevalence of this variant in a sample of prevalent prostate cancer cases managed in urology consultation in Martinique .

DETAILED DESCRIPTION:
In Martinique, prostate cancer incidence rates are nowadays among the highest worldwide with a high incidence of early-onset and familial forms. Despite the demonstration of a strong familial component, identification of the genetic basis for hereditary prostate cancer is challenging. The screening of the HOXB13 gene is recommended for men who develop an early-onset and/or familial Pca . In fact, the HOXB13 germline variant G84E (rs138213197) was described in men of European descent with prostate cancer risk. Other germline variants were detected in ethnic groups. More recently, we reported a rare HOXB13 mutation, specifically c.853delT (pTer285Lysfs) that appears to be contribute to young Prostate Cancer cases in Martinique. This variant is a stop loss reported only among patients of African ancestry .

Regarding the allele frequency of the HOXB13 c.853delT variant observed in the Pca cohort, it will be necessary to assess relative and absolute Pca risks for HOXB13 c.853delT carriers. This information is essential to use this variant in genetic counseling. We propose to sequence the HOXB13 gene of all prostate cancers cases managed in urology consultation in Martinique.

ELIGIBILITY:
Inclusion Criteria:

* Adult man over 18 years of age living in Martinique with a prostate cancer whatever the histological type and the stage, managed in urology consultation (public and private sectors of Martinique)
* Sporadic or familial form
* Informed with a written consent signed by the participant and the investigator
* Affiliate or beneficiary of french social security.

Exclusion Criteria:

* Patient who is not of African descent
* Refusal to participate.
* Patients not affiliated to french social security

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Estimated)
Dates: Start 2021-04-09 (Actual); Primary Completion 2025-04-09 (Estimated); Study Completion 2025-04-09 (Estimated)

PRIMARY OUTCOMES:
Estimation of prevalence of Allelic frequency of the HOXB13 c.853delT mutation | At baseline
  Mutation is detected using Next Generation Sequencing (NGS) technique

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No